CLINICAL TRIAL: NCT01157806
Title: Palliative Radiotherapy Followed by Chemotherapy Against Palliative Surgery in Patients With Rectal Cancer With Unresectable Synchronous Distant Metastases
Brief Title: Palliative Radiochemotherapy Against Palliative Surgery in Stage IV Rectal Cancer With Unresectable Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Prof. Krzysztof Bujko, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology in Warsaw
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0109
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; unresectable synchronous metastases; pelvic radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiochemotherapy instead of surgery (Experimental)
  Interventions: Radiation: short course of palliative radiotherapy

INTERVENTIONS:
Radiation: short course of palliative radiotherapy — 5x5 Gy + XELOX 7 days after radiotherapy

SUMMARY:
Short course palliative radiotherapy (5x5Gy)to the pelvis in patients with symptomatic rectal tumours and with unresectable metastases may prevent palliative surgery with a good palliative outcome.The consolidating chemotherapy of XELOX may increase the efficacy of irradiation.

DETAILED DESCRIPTION:
Patients with symptomatic rectal cancer and unresectable metastases receive 25 Gy in 5 fractions of 5 Gy over 5 days to the pelvis and XELOX consolidating chemotherapy after one week. Investigators arbitrarily assumed that palliative radiotherapy to the pelvis can replace the immediate surgery if at least 30% of patients would avoid delayed surgery until the end of their lives, or for at least 18 months in the case of long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary carcinoma of the rectum (Lower border of tumour ≤ 10 cm from anal verge)
* Occurrence of subjective clinical symptoms of the primary tumor
* Non-resectable synchronous distant metastases. The decision of non-resectable metastases will be made at multidisciplinary clinical meetings.

Exclusion Criteria:

* Obstruction of the gastrointestinal tract
* Previously constructed stoma
* prior radiotherapy of the pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
percentage of patients not requiring palliative surgery during the follow-up | every three months

SECONDARY OUTCOMES:
The rate of early toxicity of radiotherapy according to the NCI CTCAE (version 3.0) | 3 months
  Assess prospectively by filling forms.
Palliative effect of radiotherapy | every three months
  Assessment of radiochemotherpy effectivenes by patients using questionaire.
Time from palliative radiotherapy to delayed palliative surgery | 18 months
Determination of prognostic factors indicating the need for immediate palliative surgery. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bujko, Prof., Principal Investigator — M. Sklodowska-Curie Memorial Cancer Centre Warsaw, Poland
Locations (1):
- M. Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland

REFERENCES:
- [Derived] Tyc-Szczepaniak D, Wyrwicz L, Kepka L, Michalski W, Olszyna-Serementa M, Palucki J, Pietrzak L, Rutkowski A, Bujko K. Palliative radiotherapy and chemotherapy instead of surgery in symptomatic rectal cancer with synchronous unresectable metastases: a phase II study. Ann Oncol. 2013 Nov;24(11):2829-34. doi: 10.1093/annonc/mdt363. Epub 2013 Sep 6. PMID 24013512